CLINICAL TRIAL: NCT03807609
Title: Does Exercise Timing Modify Post-exercise Energy Intake in Adolescents With Obesity
Brief Title: Energy Intake and Exercise Timing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Tza Nou - Maison médicale pour enfants et adolescentes - 230, rue Vercingétorix - B.P. 77 - 63150 La Bourboule (Unknown); SSR Nutrition-Obésité - 33-35 rue Maréchal Leclerc - 63000 Clermont-Ferrand (Unknown); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CHU-419
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Pediatric Obesity
Keywords: appetite control; obesity; Adolescents; exercise timing
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Exercise

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CON . (Experimental): The adolescents will be asked to remain quiet and at rest during the morning and will receive an ad libitum meal at lunch and dinner times. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
  Interventions: Other: CON . control condition without exercise / rest condition
- EX -30. (Experimental): The adolescents will be asked to complete a 30 minutes exercise set at 65% of their capacities (cycling), 30 minutes before lunch. Lunch will be served ad libitum as well as diner. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
  Interventions: Other: EX -30. Condition with an acute exercise set 30 minutes before lunch
- EX-180 (Experimental): The adolescents will be asked to complete a 30 minutes exercise set at 65% of their capacities (cycling), 30 minutes before lunch. Lunch will be served ad libitum as well as diner. Their appetite feelings will be assessed at regular intervals.
  Interventions: Other: EX-180. condition with an acute exercise set 180 minutes before lunch

INTERVENTIONS:
Other: CON . control condition without exercise / rest condition — Control condition without exercise / rest condition. The adolescents will be asked to remain quiet and at rest during the morning and will receive an ad libitum meal at lunch and dinner times. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
  Arms: CON .
Other: EX -30. Condition with an acute exercise set 30 minutes before lunch — The adolescents will be asked to complete a 30 minutes exercise set at 65% of their capacities (cycling), 30 minutes before lunch. Lunch will be served ad libitum as well as diner. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
  Arms: EX -30.
Other: EX-180. condition with an acute exercise set 180 minutes before lunch — The adolescents will be asked to complete a 30 minutes exercise set at 65% of their capacities (cycling), 30 minutes before lunch. Lunch will be served ad libitum as well as diner. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
  Arms: EX-180

SUMMARY:
The aim of the present study is to compare the effect of an exercise performed 180 or 30 minutes before lunch on the energy intake of adolescents with obesity.

DETAILED DESCRIPTION:
The present study will compare the nutritional response to the realisation of an acute exercise 180 or 30 minutes before an ad libitum buffet meal in adolescents with obesity. 18 adolescents with obesity will be asked to randomly complete three experimental sessions: i) one control session (rest); ii) one session with an acute exercise realized 180 minutes before lunch; iii) one session with the same exercise performed 30 minutes before lunch. Their ad libitum energy intake will be assessed during lunch as well as at dinner time. Appetite feelings will be assessed at regular intervals and their food reward in response to the lunch will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* - BMI percentile > 97th percentile according to the french curves.
* ages 12-16 years old
* Signed consent form
* being registered in the national social security system
* no contraindication to physical activity

Exclusion Criteria:

* Previous surgical interventions that is considered as non-compatible with the study.
* Diabetes
* weight loss during the last 6 months
* cardiovascular disease or risks

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Energy intake measured during an ad libitum buffet meal (in kcal). | at day 1
  food intake will be measured ad libitum during a lunch buffet. The adolescents will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be weighted using an electronic food scale (Casio Scale, units: grams) by a member of the investigation team and then analysed using Bilnuts software.

SECONDARY OUTCOMES:
Hunger feelings | at day 1
  hunger area under the curve will be assessed using visual analogue scale (VAS) through a the day ranging from 0 to 150, 0 being "not at all", 150 being "completely". The question asked being: How hungry are you right now?"
Food reward | at day 1
  Leeds Food Preference Questionnaire; LFPQ.Briefly, the LFPQ provides measures of the wanting and liking for an array of food images, varying in both fat content and taste.To measure the explicit liking and explicit wanting, participants are asked to rate the extent to which they "liked" or "wanted" each randomly presented food item with a 100-mm visual analogue scale. . The construct from the scales are : Explicit liking; Explicit Wanting; Implicit liking, implicit wanting, Fat Choice and Fat Taste. Each component ranged from -50 to +50. There is no total score.

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moore H, Pereira B, Fillon A, Miguet M, Masurier J, Beaulieu K, Finlayson G, Thivel D. The association between obesity severity and food reward in adolescents with obesity: a one-stage individual participant data meta-analysis. Eur J Nutr. 2024 Jun;63(4):1241-1255. doi: 10.1007/s00394-024-03348-4. Epub 2024 Feb 20. PMID 38376518
- [Derived] Fillon A, Mathieu ME, Masurier J, Roche J, Miguet M, Khammassi M, Finlayson G, Beaulieu K, Pereira B, Duclos M, Boirie Y, Thivel D. Effect of exercise-meal timing on energy intake, appetite and food reward in adolescents with obesity: The TIMEX study. Appetite. 2020 Mar 1;146:104506. doi: 10.1016/j.appet.2019.104506. Epub 2019 Oct 31. PMID 31678149